CLINICAL TRIAL: NCT06849466
Title: Effect of Perioperative Dexmedetomidine Sleep Promotion Management on Chronic Post-Surgical Pain: A Randomized Controlled Trial
Brief Title: Effect of Perioperative Dexmedetomidine on Chronic Post-Surgical Pain
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: National Cancer Center/National Cancer Clinical Medical Research Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College (Unknown)
Responsible Party: Principal Investigator, Lu Che, Attending Anesthesiologist, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: K7581
Record Dates: First submitted 2025-02-17; First posted 2025-02-27 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Chronic Post-Surgical Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine group (Experimental): Patients in the dexmedetomidine group will receive intranasal dexmedetomidine from 1 day before surgery until 1 day prior to discharge. After being instructed on the usage method by the research team, patients will be guided to self-administer the dexmedetomidine nasal spray between 21:00 and 21:30.
  The dosage will be based on body weight and will be as follows:
  For patients weighing 40-49 kg: 2 sprays (50 µg) For patients weighing 50-69 kg: 3 sprays (75 µg) For patients weighing 70-89 kg: 4 sprays (100 µg) For patients weighing 90-100 kg: 5 sprays (125 µg) After administration, patients will be instructed to lie flat and prepare for sleep. Objective sleep quality will be monitored using wearable sleep monitoring devices.
  Interventions: Drug: Dexmedetomidine
- Control group (Placebo Comparator): Patients in the control group will receive intranasal placebo from 1 day before surgery until 1 day prior to discharge. After being instructed on the usage method by the research team, patients will be guided to self-administer an equal volume of spray between 21:00 and 21:30. Patients will be instructed to use the spray while in a semi-recumbent position, with saline solution administered based on the corresponding dosage:
  For patients weighing 40-49 kg: 2 sprays For patients weighing 50-69 kg: 3 sprays For patients weighing 70-89 kg: 4 sprays For patients weighing 90-100 kg: 5 sprays After administration, patients will be instructed to lie flat and prepare for sleep. Objective sleep quality will be monitored using wearable sleep monitoring devices
  Interventions: Drug: Saline solution

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine Hydrochloride Nasal Spray Dexmedetomidine is a selective alpha-2 adrenergic agonist primarily used for its sedative, anxiolytic, and analgesic effects. It works by inhibiting the release of norepinephrine in the central nervous system, leading to sedation, decreased anxiety, and reduced pain sensitivity. When used intranasally, it can offer an effective, non-invasive method for sedating patients and improving sleep quality, particularly in perioperative settings.
  Arms: Dexmedetomidine group
Drug: Saline solution — The saline solution will be used as a placebo, and the same device will be employed for intranasal administration.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn if intranasal dexmedetomidine works to improve sleep quality to treat chronic post-surgical pain (CPSP) in patients undergoing thoracic surgery. It will also learn about the safety of intranasal dexmedetomidine.this clinical trial could include any of the following: Adults aged 18-80 years, Elective surgical patients scheduled for their first thoracoscopic lung resectiony, ASA physical status I-III, and sign the informed consent form. The main questions it aims to answer are:

Does intranasal dexmedetomidine reduce the incidence of CPSP in patients undergoing elective thoracic surgery? Does perioperative sleep quality mediates the effect of intranasal dexmedetomidine in improving CPSP outcomes at 3 months post-surgery? What are the safety concerns or medical complications that participants may experience when using intranasal dexmedetomidine perioperatively? Researchers will compare the intervention group receiving intranasal dexmedetomidine to a placebo (a look-alike substance that contains no drug) to assess its impact on perioperative sleep quality and the reduction in CPSP incidence at 3 months post-surgery.

Participants will:

Take the study drug (intranasal dexmedetomidine) or a placebo (saline) every night between 9:00-9:30 PM, starting the day before surgery and continuing until the day before discharge.

After the drug administration, undergo 3 hours of continuous monitoring with ECG and wear a wearable device for ongoing assessment.

Cooperate with researchers to assess sedation, pain, sleep, emotional status, medication usage, adverse events, and postoperative recovery quality on postoperative days 1, 2, and 3 You will be contacted by phone at 1, 3, and 6 months by the research team to inquire about sleep, pain, medication use, and overall quality of life after discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-80 years,
2. Elective surgical patients scheduled for their first thoracoscopic lung resectiony,
3. ASA physical status I-III
4. sign the informed consent form

Exclusion Criteria:

1. Severe heart failure or left ventricular ejection fraction (LVEF) <30%, or the presence of coronary artery disease, cardiac conduction abnormalities, or arrhythmias;
2. Abnormal liver function, defined as ALT >100 IU/L or Child-Pugh Class B;
3. Renal insufficiency, characterized by an estimated glomerular filtration rate (eGFR) <60 mL/min or a preoperative serum creatinine level >120 µmol/L;
4. A history of peptic ulcer disease, gastrointestinal bleeding, asthma, or cerebrovascular disease;
5. Known allergy to medications potentially used in this study, including dexmedetomidine, propofol, opioids, nonsteroidal anti-inflammatory drugs (NSAIDs), or local anesthetics;
6. Body mass index (BMI) >30 kg/m²;
7. Preoperatively diagnosed psychiatric disorders, such as anxiety, depression, or sleep disturbances;
8. Long-term use of opioids or sedatives, defined as usage for 3 months or longer;
9. Pregnant women, postpartum individuals, and breastfeeding mothers;
10. Patients anticipated to require postoperative admission to the intensive care unit (ICU);
11. Patients with nasal abnormalities or conditions that preclude or contraindicate intranasal drug administration.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of chronic post-surgical pain (CPSP): Brief Pain Inventory (BPI) and Douleur Neuropathique 4 Questions (DN4） | at 3 months after surgery
  Phone interviews were conducted at 3 months after surgery by trained pain physicians following a standardized protocol at each participating centre. Primarily, the question was asked: "Do you currently have persisting pain related to your thoracoscopic surgery ?" If the answer is "YES", the BPI and DN-4 (Douleur Neuropathique4 questions, as Neuropathic pain four questions in English) were applied for pain evaluation. After that, CPSP will be finally diagnosed focusing on key diagnostic criteria including: (1) Pain arises or intensifies following surgery; (2) Pain persists for at least three months and impacts quality of life; (3) Pain occurs after a pain-free interval or evolves from ongoing acute postoperative pain; (4) Pain is localized to the surgical site or radiates to areas corresponding to the relevant nerve distribution; and (5) Other potential causes of pain have been excluded.

SECONDARY OUTCOMES:
Subjective sleep assessment: Pittsburgh Sleep Quality Index (PSQI) | 1, 3, and 6 months after surgery.
  The Pittsburgh Sleep Quality Index (PSQI), developed by Dr. Daniel J. Buysse and his colleagues at the University of Pittsburgh in 1989, contains 19 self-rated and 5 observer-rated questions grouped into 7 components including subjective sleep quality and sleep latency etc., with each component scored 0 - 3 and total score 0 - 21, where 5 or less means good sleep quality and 5 or more indicates poor sleep quality, and it's widely used in sleep medicine, psychology and clinical research to evaluate sleep problems, monitor treatment effects and conduct epidemiological investigations, being a reliable and valid tool for assessing sleep quality and crucial for understanding and managing sleep-related issues.
Subjective sleep assessment: Richards - Campbell Sleep Questionnaire (RCSQ) | 1st, 2nd, and 3rd days after surgery.
  The Richards-Campbell Sleep Questionnaire (RCSQ) is a prominent tool in sleep research and clinical practice for gauging sleep quality. It comprehensively evaluates sleep aspects from respondents' subjective views.
  Comprising multiple items, it covers sleep onset latency (time to fall asleep), sleep depth, sleep duration, and wake-up frequency at night. It may also involve related factors like sleep environment quality and sleep's impact on daily life.
  With specific questions and response options, individuals rate sleep experiences numerically or descriptively. Data from the RCSQ aids in diagnosing sleep disorders, evaluating treatment efficacy, and conducting sleep-related epidemiological studies. It is mainly intended for the assessment of short-term sleep conditions during hospitalization.
Objective sleep assessment: Total sleep duration, wake - up time during sleep, and deep sleep time. | 1st, 2nd, and 3rd days after surgery
  We will use Huawei smart wearable devices to assess the objective sleep conditions of patients. The definition of total sleep duration is as follows: Before the sleep on the first night before their surgery, a wearable sleep monitoring device was placed on the non-dominant wrist of each participant. The patients wore this sleep monitoring device throughout their hospitalization. The sleep monitoring period is from 20:00 to 20:00 the next day.
  The indicator of Wake-up time during sleep refers to the total time a person is awake after initially falling asleep.
  The deep sleep duration: According to Huawei's scientific sleep (TruSleep™) technology, the sleep status of patients is determined by analyzing data such as the patients' heart rate and body movements, and it is recorded.
Emotional state assessment: Hospital Anxiety and Depression Scale (HADS) | 1st, 2nd, and 3rd days after surgery
  The Hospital Anxiety and Depression Scale (HADS) is a widely utilized psychological assessment tool. It aims to screen and evaluate anxiety and depression levels of patients in hospital or clinical settings. Comprising 14 items split into an Anxiety Subscale and a Depression Subscale with 7 items each, it assesses symptoms related to both. Respondents rate items based on their past week's feelings. Proven reliable and valid across diverse populations and cultures, it's handy in medical settings for differentiating coexisting mental symptoms with physical illnesses. Easy to administer and score, it's crucial for early detection, treatment planning, and monitoring, aiding comprehensive mental health management.
Pain assessment: Numerical rating scale (NRS) | 1st, 2nd, 3rd days after surgery and at 1, 2, 3, 6 months after surgery
  The Numerical Rating Scale (NRS) for pain is a commonly used tool in healthcare to gauge patients' pain intensity. It's a subjective measure where patients rate pain on a 0 - 10 scale. 0 means no pain; 10 is the worst imaginable pain. Scores 3 and below suggest mild pain with little impact, 4 - 6 moderate pain affecting daily life somewhat, and 7 and above severe pain needing prompt attention.
  It's practical for its simplicity. Medical staff can administer it quickly during consultations. Patients can easily understand and use it to convey pain feelings. This helps professionals evaluate pain severity, plan treatments, and monitor pain relief. Overall, the NRS is vital in pain assessment and management, enhancing medical care quality and patient comfort.
Quality of recovery assessment: Quality of Recovery-15 (QoR-15) assessment scale | 1st and 3rd days after surgery
  The Quality of Recovery-15 (QoR-15) assessment scale is a professional tool for evaluating the recovery quality of patients post-surgery or after certain medical interventions. It is composed of 15 items, with each item scored from 0 to 10 points, and the total score ranges from 0 to 150 points. The higher the score, the better the quality of recovery.
  These 15 items cover five dimensions: physical comfort, emotional state, physical independence, psychological support, and pain. The QoR-15 scale is recognized for its high reliability and validity. It is easy to administer and score, which is of great significance in assessing patients' recovery status and guiding medical staff to formulate appropriate treatment and care plans.
Quality of life assessment: Short Form-36 Health Survey Questionnaire (SF-36) | 1, 3, 6 months after surgery
  Short Form-36 Health Survey Questionnaire (SF-36) The SF-36 is a widely recognized and commonly used instrument for assessing quality of life. It consists of 36 questions covering eight domains, such as physical functioning, role limitations due to physical problems, social functioning, and mental health.The scale provides a comprehensive view of an individual's quality of life, generating scores that help healthcare providers understand patients' well-being and make more informed decisions in diagnosis, treatment, and care, with good reliability and validity demonstrated in various studies.
Incidence of chronic post-surgical pain (CPSP) : Brief Pain Inventory (BPI) and Douleur Neuropathique 4 Questions (DN4) | at 6 months after surgery
  Phone interviews were conducted at 3 months after surgery by trained pain physicians following a standardized protocol at each participating centre. Primarily, the question was asked: "Do you currently have persisting pain related to your thoracoscopic surgery ?" If the answer is "YES", the BPI and DN-4 (Douleur Neuropathique4 questions, as Neuropathic pain four questions in English) were applied for pain evaluation. After that, CPSP will be finally diagnosed focusing on key diagnostic criteria including: (1) Pain arises or intensifies following surgery; (2) Pain persists for at least three months and impacts quality of life; (3) Pain occurs after a pain-free interval or evolves from ongoing acute postoperative pain; (4) Pain is localized to the surgical site or radiates to areas corresponding to the relevant nerve distribution; and (5) Other potential causes of pain have been excluded.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The data generated from this study are anonymized datasets with all patient-identifying information, including but not limited to names, ID numbers, contact details, and biometric features, completely removed.
Supporting Information: Study Protocol, SAP
Access Criteria: For data access, interested parties should submit a formal request to the corresponding author of this study via pumchshenle@163.com. The request must contain a detailed data usage plan, a rational justification, and clear objectives for data utilization. All data requests are subject to review by the Peking Union Medical College Hospital Institutional Review Board. Only after ethical and legal assessments confirm compliance with relevant regulations and ensure no potential risks to study participants will the data be provided to the applicants.Moreover, supplementary information such as the study protocol or statistical analysis plan can be made available concurrently upon approval of the reasonable data request. The data are only permitted for use within the boundaries of ethical and legal permissions. Secondary dissemination or utilization for other research purposes without prior written authorization is strictly prohibited.

REFERENCES:
- [Derived] Xu L, Zhang Y, Che L, Shen L. Perioperative intranasal dexmedetomidine for the prevention of chronic postsurgical pain following thoracoscopic surgery: protocol for a multicentre randomised controlled trial. BMJ Open. 2025 Aug 8;15(8):e105832. doi: 10.1136/bmjopen-2025-105832. PMID 40780715